CLINICAL TRIAL: NCT05174663
Title: A Randomized, Comparator-controlled Parallel Study to Investigate the Dose Response of an Almond-enriched Diet on Optimizing HDL-C in a Population With Hypercholesterolemia
Brief Title: Investigating the Dose Response of an Almond-enriched Diet on Optimizing HDL-C in a Population With Hypercholesterolemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Almond Board of California (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21ABCFA01
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-01

CONDITIONS: HDL-C; Hypercholesterolemia
Keywords: Hypercholesterolemia; HDL-C; Almond-enriched diet
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The dietary interventions in this proposed study prevent blinding as it is impossible to mask the participant and investigators to whether the participants are consuming whole almonds or not. The requirements to report the quantity of almonds consumed also precludes blinding for both the participant and investigator. The statistician will be blinded for the duration of the study and throughout all analysis and reporting. The preclusion of blinding in this study is not a limitation given the objectivity of the primary and most secondary endpoints. This is a well-controlled study design that provides a "real-world" assessment of the dietary interventions that bolsters the resulting data to withstand scientific and regulatory scrutiny.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Almond-enriched diet dose 1 (Experimental): Participants will be instructed to ingest 1.5 oz of almonds daily for 16 weeks. The 1.5 oz of almonds can be split into a morning and afternoon snack. Participants will be advised not to exceed 2 doses of almonds daily. If a dose is missed, participants should take the missed dose as soon as the participants remember.
  Interventions: Other: Almond-enriched diet - 1.5 oz
- Almond-enriched diet dose 2 (Experimental): Participants will be instructed to ingest 2.5 oz of almonds daily for 16 weeks. The 2.5 oz of almonds can be split into a morning and afternoon snack. Participants will be advised not to exceed 2 doses of almonds daily. If a dose is missed, participants should take the missed dose as soon as the participants remember.
  Interventions: Other: Almond-enriched diet - 2.5 oz
- Nut-free diet (Other): Participants will be instructed to ingest the control snack (Iso-caloric [to 1.5 oz of almonds] control snack of chocolate chip cookies or Oreo cookies) daily for 16 weeks. The control snack can be split into a morning and afternoon snack. Participants will be advised not to exceed 2 doses of snack daily. If a dose is missed, participants should take the missed dose as soon as the participants remember.
  Interventions: Other: Control snack

INTERVENTIONS:
Other: Almond-enriched diet - 1.5 oz — Participants will receive 1.5 oz of almonds consumed as a snack daily for 16 weeks.
  Arms: Almond-enriched diet dose 1
Other: Almond-enriched diet - 2.5 oz — Participants will receive 2.5 oz of almonds consumed as a snack daily for 16 weeks.
  Arms: Almond-enriched diet dose 2
Other: Control snack — Participants will receive a control snack daily for 16 weeks.
  Arms: Nut-free diet

SUMMARY:
This study will determine the quantity of almonds (1.5 oz or 2.5 oz) consumed as a snack that will provide optimal increases in HDL-C levels.

DETAILED DESCRIPTION:
Elevated lipid levels are a major modifiable risk factor for cardiovascular disease (CVD), which is the leading cause of death worldwide, accounting for over 17.8 million deaths globally, equating to approximately 71 million Americans with the total annual cost associated with CVD approximating $351.3 billion USD. The National Cholesterol Education Program (NCEP) ATP III Guidelines and supporting literature recommend diet and lifestyle approaches for patients with elevated lipid levels prior to lipid lowering medication, as changing lifestyle and diet cost less than medications and does not lead to polypharmacy or unwanted side effects. Low nut and seed consumption has been identified as the leading dietary risk factor attributed to ischemic heart disease. Indeed, studies have demonstrated that almond consumption reduces total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), and triglyceride (TG) levels compared to no almond controls or substitutions. Additionally, emerging and predictive CVD risk factors such as abdominal obesity and concentrations of Apolipoprotein (ApoB), for which a dose-response effect may also be present, are also improved by almond consumption.

While the benefits of an almond-rich diet on TC, TG, and LDL-C are clear, the effects of almonds on high-density lipoprotein cholesterol (HDL-C) levels is less clear. In populations with hyperlipidemia, almond consumption appears to improve HDL-C, among other lipid markers. Yet, a recent systematic-review and meta-analysis reported a significant decrease in HDL-C compared to control across 12 studies. It is possible that a dose-response relationship exists for almond consumption and HDL-C levels. Almond consumption of ≤42.5 g/day significantly decreased LDL-C/HDL-C, TC/HDL-C and ApoB compared to control, however, significant reductions in TC, BP and body weight were only observed with >42.5 g of almonds/day. Sabate et al., found that the NCEP Step I Diet as well as a low almond diet (10% from calories) significantly reduced HDL-C by 3% and 4%, respectively. However, a high almond-diet (20% from calories) maintained HDL-C levels, while having favorable changes on LDL-C, LDL-C/HDL-C and ApoB/ApoA . Daily almond consumption between 37-73 g/day (~1.3-2.5 oz/day) resulted in significantly higher HDL-C levels compared to a muffin control, with the higher dose of almonds (73 g/day) resulting in a greater increase in HDL-C compared to a lower dose (37 g/day). Additionally, the majority of studies are of limited length and often less than 12 weeks long. A previous study on the long term effects of almonds and other lipid-modulating foods found the greatest reductions on LDL-C and TC/HDL-C were not observed until 12 weeks, and then maintained. Further, it has been suggested that other outcomes such as BP, body weight and abdominal obesity may require longer term consumption of almonds to show beneficial changes. Therefore, it is likely heterogeneity in the effect of HDL-C levels with almond consumption is due to inadequate study duration, background diet, population, control used or too low quantity of almonds.

The existing FDA health claim for almonds states: "scientific evidence suggests, but does not prove, that eating 1.5 ounces per day of most nuts, such as almonds, as part of a diet low in saturated fat and cholesterol may reduce the risk of heart disease". Despite the benefits of almonds on cardiometabolic health, clinical trials designed to determine the optimal dose of almonds on the improvement of lipid profile in a population at greater risk of CVD have not been conducted. This study will address this research gap and establish the optimal dose of almonds for improving HDL-C and other CVD markers and ultimately lowering risk in a population at increased risk of disease development. The specific aim of this study is to demonstrate the efficacy of consuming increasing quantities of almonds on blood lipid levels in adults with hypercholesterolemia. Two doses of almonds will be used, 1.5 oz and 2.5 oz, referred to the Almond-enriched Diet Dose 1 (AD1) and Almond-enriched Diet Dose 2 (AD2), respectively, compared to a Nut-Free Diet (NFD). This study will determine the optimal quantity of almonds consumed as a snack that will provide the most clinically relevant increase of HDL-C levels. Further, this study will investigate the dose-response of almonds on other lipid profile markers, blood pressure (BP), weight, and markers of abdominal obesity in a population with hypercholesterolemia. The hypothesis is that there will be an improvement in HDL-C in a dose-dependent manner with increased consumption of almonds for 16 weeks.

Participants in this study represent a target population that aligns with the goals of healthcare to provide lifestyle management prior to the introduction of prescription medication plans. The study is to be conducted in a population at risk of developing heart disease, who have hypercholesterolemia based on the NCEP definition (LDL-C levels >4.1 mmol/L (>160 mg/dL)). Currently, approximately 53% of the North American population is considered to have elevated LDL-C levels, yet less than half receive treatment. Participants aged 30 to 65 years will be considered for enrolment to avoid complications related to advanced age and a body mass index (BMI) of and up to 34.9 kg/m2 will eliminate confounders related to advanced obesity. Significant metabolic or physiological conditions that may affect lipid levels will be excluded and any participants on prescribed lipid lowering medication will be excluded to limit confounders. Current use of supplements known to affect blood lipid levels, vitamin E status or tree nuts that may impact study outcomes will be excluded unless participants undergo an appropriate washout period prior to enrollment. As well, an extensive list of exclusions in place will ensure that eligibility is based on establishing health and each participants' eligibility will be overseen by the Qualified Investigator (QI).

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females between 30-65 years of age, inclusive
2. BMI between 25.0 - 34.9 kg/m2, inclusive
3. Individual is not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
4. Individuals with hypercholesterolemia based on the NCEP definition (LDL-C levels >4.1 mmol/L (>160 mg/dL))
5. Motivated to comply with dietary guidelines as assessed by a motivation questionnaire at screening
6. Self-reported stable body weight for the past 3 months defined as not having gained or lost more than 5 kg of body weight throughout the 3 months prior to baseline
7. Agrees to adhere to dietary guidelines and to maintain current lifestyle habits as much as possible throughout the study depending on the participants' ability to maintain the following: medications, supplements, exercise, and sleep and avoid taking new supplements
8. Provided voluntary, written, informed consent to participate in the study
9. Healthy as determined by medical history, and laboratory results exam as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product/control snack ingredients
3. Current regular consumption of nuts >2 times per week, unless willing to washout prior to baseline
4. Current use of prescribed lipid lowering medications as assessed by QI (see Section 7.3.1)
5. Current use of over-the-counter medications or supplements known to affect blood lipid levels (i.e. omega-3) or vitamin E status
6. Unstable metabolic disease or chronic diseases as assessed by the QI
7. Current or history of any significant diseases of the gastrointestinal tract as assessed by QI
8. Type I or Type II diabetes
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Individuals with an autoimmune disease or are immune compromised as assessed by QI
14. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis
15. Self-reported confirmation of blood/bleeding disorders as assessed by QI
16. Use of tobacco products within 12 weeks of baseline and during the study period as assessed by QI
17. Alcohol intake average of >2 standard drinks per day as assessed by the QI
18. Alcohol or drug abuse within the last 12 months
19. Clinically significant abnormal laboratory results at screening as assessed by the QI
20. Individuals who are unable to give informed consent
21. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 16 in HDL-C levels between the Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, and Nut-Free Diet | 16 weeks
  The change from baseline in HDL-C levels at week 16 between Almond-enriched Diet Dose 1 (AD1), Almond-Enriched Diet Dose 2 (AD2), and Nut-Free Diet (NFD) will be determined.

SECONDARY OUTCOMES:
Change from baseline to week 4 in HDL-C levels between the Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, and Nut-Free Diet | 4 weeks
  The change from baseline in HDL-C levels at week 4 between Almond-enriched Diet Dose 1 (AD1), Almond-Enriched Diet Dose 2 (AD2), and Nut-Free Diet (NFD) will be determined.
Change from baseline to week 8 in HDL-C levels between the Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, and Nut-Free Diet | 8 weeks
  The change from baseline in HDL-C levels at week 8 between Almond-enriched Diet Dose 1 (AD1), Almond-Enriched Diet Dose 2 (AD2), and Nut-Free Diet (NFD) will be determined.
Change from baseline to week 12 in HDL-C levels between the Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, and Nut-Free Diet | 12 weeks
  The change from baseline in HDL-C levels at week 12 between Almond-enriched Diet Dose 1 (AD1), Almond-Enriched Diet Dose 2 (AD2), and Nut-Free Diet (NFD) will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a clinically relevant increase in HDL-C levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a clinically relevant increase in HDL-C levels defined as an increase of at least 1 mg/dL (0.026 mmol/L) will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a clinically relevant increase in HDL-C levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a clinically relevant increase in HDL-C levels defined as an increase of at least 1 mg/dL (0.026 mmol/L) will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a clinically relevant increase in HDL-C levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a clinically relevant increase in HDL-C levels defined as an increase of at least 1 mg/dL (0.026 mmol/L) will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a clinically relevant increase in HDL-C levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a clinically relevant increase in HDL-C levels defined as an increase of at least 1 mg/dL (0.026 mmol/L) will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving no change or an increase in HDL-C levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving no change or an increase in HDL-C levels based on expected effects through almond intervention will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving no change or an increase in HDL-C levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving no change or an increase in HDL-C levels based on expected effects through almond intervention will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving no change or an increase in HDL-C levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving no change or an increase in HDL-C levels based on expected effects through almond intervention will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving no change or an increase in HDL-C levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving no change or an increase in HDL-C levels based on expected effects through almond intervention will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving movement from HDL-C categories | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving movement from HDL-C categories defined by NCEP guidelines (those with HDL-C levels <40 mg/dL (1.04 mmol/L) and ≥40 mg/dL) will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving movement from HDL-C categories | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving movement from HDL-C categories defined by NCEP guidelines (those with HDL-C levels <40 mg/dL (1.04 mmol/L) and ≥40 mg/dL) will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving movement from HDL-C categories | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving movement from HDL-C categories defined by NCEP guidelines (those with HDL-C levels <40 mg/dL (1.04 mmol/L) and ≥40 mg/dL) will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving movement from HDL-C categories | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving movement from HDL-C categories defined by NCEP guidelines (those with HDL-C levels <40 mg/dL (1.04 mmol/L) and ≥40 mg/dL) will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in total cholesterol levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in total cholesterol levels will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in total cholesterol levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in total cholesterol levels will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in total cholesterol levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in total cholesterol levels will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in total cholesterol levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in total cholesterol levels will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in LDL-C levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in LDL-C levels will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in LDL-C levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in LDL-C levels will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in LDL-C levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in LDL-C levels will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in LDL-C levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in LDL-C levels will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in triglyceride levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in triglyceride levels will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in triglyceride levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in triglyceride levels will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in triglyceride levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in triglyceride levels will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in triglyceride levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in triglyceride levels will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in non-HDL-C levels | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in non-HDL-C levels will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in non-HDL-C levels | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in non-HDL-C levels will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in non-HDL-C levels | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in non-HDL-C levels will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in non-HDL-C levels | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in non-HDL-C levels will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in the Triglyceride/HDL-C ratio | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in the Triglyceride/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in the Triglyceride/HDL-C ratio | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in the Triglyceride/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in the Triglyceride/HDL-C ratio | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in the Triglyceride/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in the Triglyceride/HDL-C ratio | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in the Triglyceride/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in the Total Cholesterol/HDL-C ratio | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in the Total Cholesterol/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in the Total Cholesterol/HDL-C ratio | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in the Total Cholesterol/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in the Total Cholesterol/HDL-C ratio | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in the Total Cholesterol/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in the Total Cholesterol/HDL-C ratio | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in the Total Cholesterol/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 4 weeks achieving a change in the LDL-C/HDL-C ratio | 4 weeks
  The difference in the proportion of participants from baseline to 4 weeks achieving a change in the LDL-C/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 8 weeks achieving a change in the LDL-C/HDL-C ratio | 8 weeks
  The difference in the proportion of participants from baseline to 8 weeks achieving a change in the LDL-C/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 12 weeks achieving a change in the LDL-C/HDL-C ratio | 12 weeks
  The difference in the proportion of participants from baseline to 12 weeks achieving a change in the LDL-C/HDL-C ratio will be determined.
The difference in the proportion of participants from baseline to 16 weeks achieving a change in the LDL-C/HDL-C ratio | 16 weeks
  The difference in the proportion of participants from baseline to 16 weeks achieving a change in the LDL-C/HDL-C ratio will be determined.
The difference in change in ApoB48 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks | 8 weeks
  The difference in change in ApoB48 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks will be determined.
The difference in change in ApoB48 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks | 16 weeks
  The difference in change in ApoB48 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks will be determined.
The difference in change in ApoB100 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks | 16 weeks
  The difference in change in ApoB100 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks will be determined.
The difference in change in ApoB100 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks | 8 weeks
  The difference in change in ApoB100 concentration between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks will be determined.
The difference in change in cardiovascular disease risk between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks | 8 weeks
  The difference in change in cardiovascular disease (CVD) risk between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 8 weeks will be determined. Cardiovascular disease risk scores will be assessed by Framingham CVD Risk Scores, which is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual.
The difference in change in cardiovascular disease risk between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks | 16 weeks
  The difference in change in cardiovascular disease (CVD) risk between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet from baseline to 16 weeks will be determined. Cardiovascular disease risk scores will be assessed by Framingham CVD Risk Scores, which is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual.
The change in weight from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in weight from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in weight from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in weight from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in weight from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in weight from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in weight from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in weight from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Body Mass Index from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in Body Mass Index from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Body Mass Index from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in Body Mass Index from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Body Mass Index from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in Body Mass Index from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Body Mass Index from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in Body Mass Index from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Sagittal Abdominal Diameter from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in Sagittal Abdominal Diameter from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Also known as abdominal height, Sagittal Abdominal Diameter will be measured with the participant in a supine position with straight legs after normal expiration. At the level of the iliac crest, Sagittal Abdominal Diameter is the distance between the examination table to the horizontal level using abdominal calipers. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 0.5 cm, a third measurement is to be taken and the two closest values will be averaged for final measurement.
The change in Sagittal Abdominal Diameter from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in Sagittal Abdominal Diameter from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Also known as abdominal height, Sagittal Abdominal Diameter will be measured with the participant in a supine position with straight legs after normal expiration. At the level of the iliac crest, Sagittal Abdominal Diameter is the distance between the examination table to the horizontal level using abdominal calipers. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 0.5 cm, a third measurement is to be taken and the two closest values will be averaged for final measurement.
The change in Sagittal Abdominal Diameter from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in Sagittal Abdominal Diameter from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Also known as abdominal height, Sagittal Abdominal Diameter will be measured with the participant in a supine position with straight legs after normal expiration. At the level of the iliac crest, Sagittal Abdominal Diameter is the distance between the examination table to the horizontal level using abdominal calipers. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 0.5 cm, a third measurement is to be taken and the two closest values will be averaged for final measurement.
The change in Sagittal Abdominal Diameter from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in Sagittal Abdominal Diameter from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Also known as abdominal height, Sagittal Abdominal Diameter will be measured with the participant in a supine position with straight legs after normal expiration. At the level of the iliac crest, Sagittal Abdominal Diameter is the distance between the examination table to the horizontal level using abdominal calipers. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 0.5 cm, a third measurement is to be taken and the two closest values will be averaged for final measurement.
The change in Waist Circumference from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in Waist Circumference from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Measurements will be performed when standing at the part of the trunk located midway between the lower costal margin and the iliac crest. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 10%, a third measurement is to be taken and the two closest values will be averaged for final measurement. The height of the waist will be also recorded at baseline, and then used to determine the waist throughout the study in order to ensure a consistent measurement at all visits.
The change in Waist Circumference from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in Waist Circumference from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Measurements will be performed when standing at the part of the trunk located midway between the lower costal margin and the iliac crest. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 10%, a third measurement is to be taken and the two closest values will be averaged for final measurement. The height of the waist will be also recorded at baseline, and then used to determine the waist throughout the study in order to ensure a consistent measurement at all visits.
The change in Waist Circumference from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in Waist Circumference from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Measurements will be performed when standing at the part of the trunk located midway between the lower costal margin and the iliac crest. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 10%, a third measurement is to be taken and the two closest values will be averaged for final measurement. The height of the waist will be also recorded at baseline, and then used to determine the waist throughout the study in order to ensure a consistent measurement at all visits.
The change in Waist Circumference from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in Waist Circumference from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined. Measurements will be performed when standing at the part of the trunk located midway between the lower costal margin and the iliac crest. At least two separate measurements are to be taken at each visit. If the two measurements differ by more than 10%, a third measurement is to be taken and the two closest values will be averaged for final measurement. The height of the waist will be also recorded at baseline, and then used to determine the waist throughout the study in order to ensure a consistent measurement at all visits.
The change in Waist to Hip Ratio from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in Waist to Hip Ratio from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Waist to Hip Ratio from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in Waist to Hip Ratio from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Waist to Hip Ratio from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in Waist to Hip Ratio from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in Waist to Hip Ratio from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in Waist to Hip Ratio from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in blood pressure from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 4 weeks
  The change in blood pressure from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in blood pressure from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 8 weeks
  The change in blood pressure from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in blood pressure from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 12 weeks
  The change in blood pressure from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The change in blood pressure from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet | 16 weeks
  The change in blood pressure from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The difference in change in serum α-tocopherol concentrations from baseline to 16 weeks between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet | 16 weeks
  The difference in change in serum α-tocopherol concentrations from baseline to 16 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The difference in change in serum α-tocopherol concentrations from baseline to 12 weeks between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet | 12 weeks
  The difference in change in serum α-tocopherol concentrations from baseline to 12 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The difference in change in serum α-tocopherol concentrations from baseline to 8 weeks between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet | 8 weeks
  The difference in change in serum α-tocopherol concentrations from baseline to 8 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.
The difference in change in serum α-tocopherol concentrations from baseline to 4 weeks between Almond-enriched Diet Dose 1 and Almond-Enriched Diet Dose 2 compared to the Nut-Free Diet | 4 weeks
  The difference in change in serum α-tocopherol concentrations from baseline to 4 weeks between Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2 and the Nut-Free Diet will be determined.

OTHER OUTCOMES:
Incidence of pre-emergent adverse events following 16-week ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks and at a 7-day follow-up at the end of the study
  Incidence of pre-emergent adverse events following 16-week ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Incidence of post-emergent adverse events following 16-week ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks and at a 7-day follow-up at the end of the study
  Incidence of post-emergent adverse events following 16-week ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in Aspartate Aminotransferase levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in Aspartate Aminotransferase levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in alanine aminotransferase levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in alanine aminotransferase levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in alkaline phosphatase from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in alkaline phosphatase from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in total bilirubin levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in total bilirubin levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in creatinine from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in creatinine from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in potassium levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in potassium levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in sodium levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in sodium levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in chloride levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in chloride levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in glucose levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in glucose levels from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in estimated glomerular filtration rate (eGFR) from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in estimated glomerular filtration rate (eGFR) from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in white blood cell count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in white blood cell count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of neutrophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of neutrophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of lymphocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of lymphocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of monocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of monocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of eosinophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of eosinophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of basophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of basophils from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of hemoglobin from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of hemoglobin from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of hematocrit from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of hematocrit from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in Red Blood Cell (RBC) Count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in Red Blood Cell (RBC) Count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in platelet count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in platelet count from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of immature granulocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of immature granulocytes from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in levels of nucleated red blood cells from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in levels of nucleated red blood cells from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in mean corpuscular volume from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in mean corpuscular volume from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in mean corpuscular hemoglobin from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in mean corpuscular hemoglobin from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in mean corpuscular hemoglobin concentration from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in mean corpuscular hemoglobin concentration from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined.
Change in red cell distribution width from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet | 16 weeks
  Change in red cell distribution width from baseline to 16 weeks following daily ingestion of Almond-enriched Diet Dose 1, Almond-Enriched Diet Dose 2, or Nut-Free Diet will be determined. Red cell distribution width is expressed as a percentage of variation.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada